CLINICAL TRIAL: NCT01176032
Title: The "ALiskiren or Losartan Effects on bioMARKers of Myocardial Remodeling (ALLMARK)" Study
Brief Title: ALiskiren or Losartan Effects on bioMARKers of Myocardial Remodeling
Acronym: ALLMARK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPP100AES02; 2009-016735-36 (EudraCT Number)
Record Dates: First submitted 2010-08-02; First posted 2010-08-05 (Estimated); Results first posted 2014-07-24 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension; Left Ventricle Hypertrophy
Keywords: Aliskiren; hypertension; concentric LVH; LV remodeling; LVMI; biomarkers; PICP; CT-1; MMP-1; TIMP-1; AnxA5; Aldosterone; Essential hypertension with concentric left ventricle hypertrophy
MeSH Terms: conditions — Hypertension | interventions — aliskiren; Losartan; Amlodipine; Hydrochlorothiazide

ARMS (2):
- Aliskiren (Experimental): Aliskiren 150 mg od for 2 weeks and up-titration to aliskiren 300 mg od for 34 weeks. In addition to the study medication, amlodipine 5mg was given to patients who did not achieve the required blood pressure (<140/90 mmHg) after 8 weeks of treatment at the maximum doses of study medication. At week 18 the dose of amlodipine was increased to 10mg if the required level (<140/90 mmHg) was still not achieved.
  HCTZ 12.5mg was prescribed at week 26 if the required values (<140/90 mmHg) had not been reached.
  Interventions: Drug: Aliskiren; Drug: Amlodipine; Drug: Hydrochlorothiazide (HCTZ)
- Lostaran (Active Comparator): Losartan 50 mg od for 2 weeks and up-titration to losartan 100 mg od for 34 weeks. In addition to the study medication, amlodipine 5mg was given to patients who did not achieve the required blood pressure (<140/90 mmHg) after 8 weeks of treatment at the maximum doses of study medication. At week 18 the dose of amlodipine was increased to 10mg if the required level (<140/90 mmHg) was still not achieved.
  HCTZ 12.5mg was prescribed at week 26 if the required values (<140/90 mmHg) had not been reached.
  Interventions: Drug: Losartan; Drug: Amlodipine; Drug: Hydrochlorothiazide (HCTZ)

INTERVENTIONS:
Drug: Aliskiren — Aliskiren 300 mg film coated tablets
  Other Names: Rasilez
  Arms: Aliskiren
Drug: Losartan — Losartan 100 mg tablets
  Arms: Lostaran
Drug: Amlodipine — Amlodipine 5mg was given to patients who did not achieve the required blood pressure (<140/90 mmHg) after 8 weeks (visit 3)of treatment at the maximum doses of study medication in addition to the study medication in order to reach the required BP. at visit 4 (week 18) the dose of amlodipine was increased to 10mg if the required level (<140/90 mmHg) was still not achieved.
Drug: Hydrochlorothiazide (HCTZ) — HCTZ 12.5mg was prescribed at visit 5 (week 26) if the required values (<140/90 mmHg) had not been reached.

SUMMARY:
The purpose of this study is to assess efficacy of aliskiren for reducing circulating levels of biomarkers of left ventricular (LV) remodeling associated with LV hypertrophy (LVH) in hypertensive patients.

DETAILED DESCRIPTION:
Blood pressure was measured 10 weeks after starting treatment (visit 3). All patients who did not achieve the required blood pressure (<140/90 mmHg) after 8 weeks of treatment at the maximum doses of study medication were given 5 mg of amlodipine in addition to the study medication in order to reach the required BP (<140/90 mmHg).

The patient's blood pressure was assessed at visit 4 (week 18) and if it was still not at the required level (<140/90 mmHg), the dose of amlodipine was increased to 10 mg.

Blood pressure was again assessed at visit 5 (week 26) and if the required values had not been reached (<140/90 mmHg), a 12.5 mg dose of hydrochlorothiazide (HCTZ) was prescribed

ELIGIBILITY:
Inclusion Criteria:

* Patient with hypertension
* Confirmed concentric left ventricular hypertrophy:
* LVMI > 49.2 g/m2.7 for men and >46.7 g/m2.7 for women
* Relative wall thickness > 0.42

Exclusion Criteria:

* Sever or secondary HTN
* LV ejection fraction of <40%
* Patient with compelling indication to ACEIs or ARBs or BB
* History of myocardial infarction, coronary artery bypass surgery, PTC intervention, TIA or stroke within 6 months of study entry
* History of collagenopathies, osteopathy
* eGFR <30 ml/min/1,73 m2, serum potassium ≥5,2 mEq/L
* Morbid obesity (BMI ≥ 42 kg/m2
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (19):
- Spain (19):
  - Novartis Investigative Site, Sanlúcar de Barrameda, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Utrera, Andalusia
  - Novartis Investigative Site, Barcelona, Barcelona
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Galdakano, Basque Country
  - Novartis Investigative Site, Vitoria-Gasteiz, Basque Country
  - Novartis Investigative Site, Burgos, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Girona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Santa Coloma de Gramanet, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Torrevieja (Alicante), Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Santander

RESULTS

PARTICIPANT FLOW:
Groups:
- Aliskiren: Aliskiren 150 mg od for 2 weeks and up-titration to aliskiren 300 mg od for 34 weeks
- Lostaran: Losartan 50 mg od for 2 weeks and up-titration to losartan 100 mg od for 34 weeks
Period: Overall Study
Arm/Group | Aliskiren | Lostaran
Started | 37 ("Started" indicates randomized and safety population) | 37
Intention-to-treat (ITT) Population | 32 | 37
Completed | 31 | 36
Not Completed | 6 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Unsatisfactory therapeutic effect | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Informed consent withdrawn | 3 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren | Lostaran | Total
Number analyzed (Participants) | 32 | 37 | 69
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.34 (9.34) | 58.05 (10.34) | 59.12 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 23 | 26 | 49

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in C-terminal Propeptide of Procollagen Type I (PICP)
Description: PICP is a measure of blood concentration of procollagen I carboxy-terminal propeptide (PICP), a peptide released from the myocardium when procollagen is converted to type I collagen. This biomarker exhibits good specificity and sensitivity for identifying myocardial fibrosis in hypertension.
Time Frame: Baseline, Week 36
Population: Intention-to-treat (ITT) population included all patients included in the safety population who had a baseline assessment of the primary variable and at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: ug/l
Arm/Group | Aliskiren | Lostaran
Number analyzed (Participants) | 32 | 37
ug/l | -5.22 (20.37) | -4.25 (24.80)

2. Secondary Outcome: Change From Baseline in Biomarkers in Heart Disease
Description: The plasma level of biomarkers parameters used to measure improvement in left ventricular (LV) function or reduction in left ventricular mass index (LVMI). The following biomarkers were analyzed: cardiotrophin-1 (CT-1), matrix metalloproteinase-1 (MMP-1); tissue inhibitor of MMPs (TIMP-1); annexin A5 (AnxA5); N-terminal prohormone of B-type natriuretic peptide (NT-proBNP)
Time Frame: Baseline, Week 36
Population: Intention-to-treat (ITT) population included all patients included in the safety population who had a baseline assessment of the primary variable and at least one post-baseline assessment. Patients with both baseline and week 36 assessment were included in this analysis.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Aliskiren | Lostaran
Number analyzed (Participants) | 32 | 37
ng/ml
  cardiotrophin-1 (CT-1) (n=32,37) | -169.15 (561.51) | -128.23 (568.02)
  matrix metalloproteinase-1 (MMP-1) (n=32,37) | 5.93 (13.33) | 5.51 (9.58)
  tissue inhibitor of MMPs (TIMP-1) (n=32,37) | -0.70 (59.18) | 9.15 (42.58)
  annexin A5 (AnxA5) (n=31,37) | -0.98 (7.33) | -1.21 (4.75)
  NT-proBNP (n=31,34) | 18.66 (165.21) | -7.55 (38.11)

3. Secondary Outcome: Change From Baseline in Biomarker Such as Aldosterone (Aldo) in Heart Disease
Description: The plasma level of biomarker parameter (aldosterone (Aldo)) used to measure improvement in left ventricular (LV) function or reduction in left ventricular mass index (LVMI)
Time Frame: Baseline, Week 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/dl
Arm/Group | Aliskiren | Lostaran
Number analyzed (Participants) | 32 | 37
ng/dl | -1.81 (27.78) | -7.90 (76.35)

4. Secondary Outcome: Change From Baseline in Left Ventricular (LV) Function, LV End-diastolic Volume by Simpson's Rule, and LV End-systolic Volume by Simpson's Rule
Description: Reductions in the following measurements were analysed between the baseline visit and the final visit: LV end-diastolic volume by Simpson's rule, and LV end-systolic volume by Simpson's rule
Time Frame: Baseline, Week 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Aliskiren | Lostaran
Number analyzed (Participants) | 32 | 37
ml
  LV end-diastolic volume (n=22,34) | 2.30 (35.65) | 0.54 (33.19)
  LV end-systolic volume (n=22,34) | -0.92 (12.24) | 0.64 (21.01)

5. Secondary Outcome: Change From Baseline in Left Ventricular (LV) Function, LV Ejection Fraction (Teicholz), and LV Ejection Fraction (Simpson)
Description: Reductions in the following measurements were analysed between the baseline visit and the final visit: LV ejection fraction (Teicholz), and LV ejection fraction (Simpson)
Time Frame: Baseline, Week 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Aliskiren | Lostaran
Number analyzed (Participants) | 32 | 37
Percent
  LV ejection fraction Teicholz(n=29,36) | 0.00 (0.11) | 0.01 (0.08)
  LV ejection fraction Simpson(n=22,34) | 0.02 (0.14) | 0.00 (0.11)

6. Secondary Outcome: Change From Baseline in Left Ventricular (LV) Function, LA (Left Atrium) Diameter
Description: Reductions in the following measurements were analysed between the baseline visit and the final visit: LA diameter
Time Frame: Baseline, Week 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm/m^2
Arm/Group | Aliskiren | Lostaran
Number analyzed (Participants) | 24 | 30
mm/m^2 | -0.13 (1.17) | -0.22 (0.98)

7. Secondary Outcome: Change From Baseline in Left Ventricular (LV) Function, Left Atrial Volume (Biplane Simpson's Method)
Description: Reductions in the following measurements were analysed between the baseline visit and the final visit: left atrial volume (biplane Simpson's method)
Time Frame: Baseline, Week 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm3/m^2
Arm/Group | Aliskiren | Lostaran
Number analyzed (Participants) | 12 | 22
cm3/m^2 | -0.55 (17.94) | -2.27 (26.46)

8. Secondary Outcome: Change From Baseline in Reduction of Left Ventricular Mass Index (LVMI)
Description: Echocardiogram was performed at week 1 and at week 36. Reduction in LVMI is defined as the difference between the LVMI at the final visit and the baseline LVMI
Time Frame: Baseline, Week 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/m^2
Arm/Group | Aliskiren | Lostaran
Number analyzed (Participants) | 32 | 37
g/m^2 | -8.05 (18.98) | -7.96 (18.69)

9. Secondary Outcome: Change From Baseline in Combination of Aliskiren With Amlodipine in Biomarkers of Heart Disease.
Description: as for outcome 2
Time Frame: Baseline, Week 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Aliskiren + Amlodipine; Losartan + Amlodipine: 5 mg of amlodipine in addition to the study medication in order to reach the required BP (<140/90 mmHg). At week 18 the dose of amlodipine can be increased to 10mg if the required level (<140/90 mmHg) was still not achieved.
- Losartan: Losartan 50 mg od for 2 weeks and up-titration to losartan 100 mg od for 34 weeks
Arm/Group | Aliskiren | Aliskiren + Amlodipine | Losartan | Losartan + Amlodipine
Number analyzed (Participants) | 15 | 17 | 16 | 21
ng/ml
  CT-1(n=15,17,16,21) | -289.18 (608.91) | -63.23 (510.91) | 156.89 (599.29) | -345.47 (443.63)
  ANXA5 (n=15,16,16,21) | -1.24 (3.70) | -0.74 (9.73) | -1.73 (4.21) | -0.81 (5.20)
  MMP-1(n=15,17,16,21) | 7.00 (10.28) | 4.99 (15.80) | 5.47 (7.88) | 5.54 (10.89)
  TIMP-1 (n=15,17,16,21) | -10.01 (73.00) | 7.51 (44.38) | 21.38 (38.40) | -0.16 (44.13)
  NT-proBNP (n=15,16,15,19) | 21.00 (214.06) | 16.46 (108.69) | -3.68 (23.78) | -10.60 (46.91)

10. Secondary Outcome: Change From Baseline in Biomarker Such as Aldosterone (Aldo) in Heart Disease in Combination of Aliskiren With Amlodipine
Description: The plasma level of biomarker parameter plasma aldosterone used to measure improvement in left ventricular (LV) function or reduction in left ventricular mass index (LVMI).
Time Frame: Baseline, Week 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/dl
Arm/Group | Aliskiren | Aliskiren + Amlodipine | Losartan | Losartan + Amlodipine
Number analyzed (Participants) | 15 | 17 | 16 | 21
ng/dl | 2.81 (21.36) | -5.89 (32.54) | -3.12 (32.45) | -11.55 (98.35)

11. Secondary Outcome: Change From Baseline in Left Ventricular (LV) Function, LV End-diastolic Volume by Simpson's Rule, and LV End-systolic Volume by Simpson's Rule in Combination of Aliskiren With Amlodipine
Description: as for outcome 4
Time Frame: Baseline, Week 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ml
Groups:
- Aliskiren + Amlodipinet; Losartan + Amlodipine: 5 mg of amlodipine in addition to the study medication in order to reach the required BP (<140/90 mmHg). At week 18 the dose of amlodipine can be increased to 10mg if the required level (<140/90 mmHg) was still not achieved.
Arm/Group | Aliskiren | Aliskiren + Amlodipinet | Losartan | Losartan + Amlodipine
Number analyzed (Participants) | 15 | 17 | 16 | 21
ml
  LV end-diastolic volume (n=11,11,15,19) | 6.60 (40.43) | -2.00 (31.51) | 5.01 (38.15) | -2.98 (29.30)
  LV end-systolic volume (n=11,11, 15,19) | -2.93 (13.24) | 1.09 (11.44) | 6.11 (23.82) | -3.69 (17.97)

12. Secondary Outcome: Change From Baseline in Left Ventricular (LV) Function, LV Ejection Fraction (Teicholz), and LV Ejection Fraction (Simpson) in Combination of Aliskiren With Amlodipine
Description: as for outcome 5
Time Frame: Baseline, Week 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Aliskiren | Aliskiren + Amlodipinet | Losartan | Losartan + Amlodipine
Number analyzed (Participants) | 15 | 17 | 16 | 21
Percent
  LV ejection fraction Teicholz (n=14,15,16,20) | 0.00 (0.09) | -0.00 (0.13) | -0.00 (0.07) | 0.01 (0.09)
  LV ejection fraction Simpson(n=11,11,15,19) | 0.05 (0.10) | -0.01 (0.17) | -0.02 (0.12) | 0.02 (0.11)

13. Secondary Outcome: Change From Baseline in Left Ventricular (LV) Function, LA (Left Atrium) Diameter in Combination of Aliskiren With Amlodipine
Description: Reductions in the following measurements were analysed between the baseline visit and the final visit: LA diameter
Time Frame: Baseline, Week 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm/m^2
Arm/Group | Aliskiren | Aliskiren + Amlodipinet | Losartan | Losartan + Amlodipine
Number analyzed (Participants) | 12 | 12 | 13 | 17
mm/m^2 | -0.18 (1.12) | -0.07 (1.27) | -0.19 (0.96) | -0.24 (1.03)

14. Secondary Outcome: Change From Baseline in Left Ventricular (LV) Function, Left Atrial Volume (Biplane Simpson's Method) in Combination of Aliskiren With Amlodipine
Description: as for outcome 7
Time Frame: Baseline, Week 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm3/m^2
Arm/Group | Aliskiren | Aliskiren + Amlodipinet | Losartan | Losartan + Amlodipine
Number analyzed (Participants) | 6 | 6 | 9 | 13
cm3/m^2 | -8.88 (15.74) | 7.78 (17.14) | -7.42 (24.37) | 1.30 (28.21)

15. Secondary Outcome: Change From Baseline of LVMI in Combination of Aliskiren With Amlodipine
Description: as for outcome 8
Time Frame: Baseline, Week 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/m2
Arm/Group | Aliskiren | Aliskiren + Amlodipinet | Losartan | Losartan + Amlodipine
Number analyzed (Participants) | 14 | 15 | 16 | 20
g/m2 | -5.68 (18.95) | -10.26 (19.40) | -3.59 (13.46) | -11.46 (21.71)

16. Secondary Outcome: Effectivness of Aliskiren in Controlling Blood Pressure Compare to Losartan in Terms of Reduction in Systolic Blood Pressure (SBP)
Description: The mean systolic BP (SBP) and diastolic BP (DBP) readings for the aliskiren and losartan treatment groups, the difference in these values between the two groups and the comparison of post-baseline vs. baseline values
Time Frame: Baseline, Week 10,18,26,36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Aliskiren | Lostaran
Number analyzed (Participants) | 32 | 37
mmHg
  Baseline, Week 10 (n=30,37) | -5.56 (12.89) | -4.03 (16.93)
  Baseline, Week 18 (n=29,36) | -9.77 (12.25) | -8.44 (17.30)
  Baseline, Week 26 (n=29,36) | -12.69 (15.05) | -10.40 (15.74)
  Baseline, Week 36 (n=32,37) | -8.87 (19.26) | -8.88 (15.91)

17. Secondary Outcome: Effectivness of Aliskiren in Controlling Blood Pressure Compare to Losartan in Terms of Reduction in Diastolic Blood Pressure (DBP)
Description: as for outcome 16
Time Frame: Baseline, Week 10,18,26,36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Aliskiren | Lostaran
Number analyzed (Participants) | 32 | 37
mmHg
  Baseline, Week 10 (n=30,37) | -1.77 (10.22) | -3.15 (10.97)
  Baseline, Week 18 (n=29,36) | -5.34 (10.66) | -7.07 (9.98)
  Baseline, Week 26 (n=29,36) | -5.34 (11.37) | -6.94 (10.10)
  Baseline, Week 36 (n=32,37) | -4.19 (10.32) | -6.68 (9.66)

18. Secondary Outcome: Effectivness of Aliskiren in Controlling Blood Pressure Compare to Losartan in Terms of Patients With Satisfactory Response Rate
Description: Response rate was defined as the proportion of patients with a satisfactory systolic BP response (SBP < 140 mmHg or reduction of ≥ 10 mmHg compared to baseline) and a satisfactory diastolic BP response (DBP < 90 mmHg or reduction of ≥ 5 mmHg compared to baseline)
Time Frame: Baseline, Week10,18,26,36
Population: as for outcome 1
Measure: Number; unit: Patients
Arm/Group | Aliskiren | Lostaran
Number analyzed (Participants) | 32 | 37
Patients
  Baseline, Week 10 | 16 | 15
  Baseline, Week 18 | 24 | 21
  Baseline, Week 26 | 24 | 27
  Baseline, Week 36 | 22 | 25

19. Secondary Outcome: Effectivness of Aliskiren in Controlling Blood Pressure Compare to Losartan in Terms of Patients With SBP < 140 mmHg and DBP < 90 mmHg Compared to Baseline
Description: The control rate was defined as the proportion of patients with SBP < 140 mmHg and DBP < 90 mmHg compared to baseline
Time Frame: Week10,18,26,36
Population: as for outcome 1
Measure: Number; unit: Patients
Arm/Group | Aliskiren | Lostaran
Number analyzed (Participants) | 32 | 37
Patients
  Control rate at Week 10 | 15 | 13
  Control rate at Week 18 | 20 | 19
  Control rate at Week 26 | 22 | 23
  Control rate at Week 36 | 21 | 20

20. Secondary Outcome: Effectivness of Aliskiren in Controlling Blood Pressure Compare to Losartan in Terms of Rate of Use of Added Antihypertensive Rescue Drugs
Description: The rate of use of first and second antihypertensive rescue drugs added was also assessed at all visits after week 2. The rescue drug at week 10 and 18 for those patients not achieving the required BP was amlodipine, Patients who did not achieve the required BP at week 26 were treated with hydrochlorothiazide
Time Frame: Baseline, Week 10,18,26
Population: as for outcome 1
Measure: Number; unit: Patients
Arm/Group | Aliskiren | Lostaran
Number analyzed (Participants) | 32 | 37
Patients
  Baseline, Week 10 (amlodipine) | 11 | 15
  Baseline, Week 18 (amlodipine) | 2 | 9
  Baseline, Week 26 (hydrochlorothiazide) | 2 | 4

ADVERSE EVENTS:
Arm/Group | Aliskiren | Losartan
Serious Adverse Events (participants affected / at risk) | 2/37 | 0/37
Other Adverse Events (participants affected / at risk) | 12/37 | 16/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren (N=37) | Losartan (N=37)
Bronchopneumonia (Infections and infestations) | 1 | 0
Coronary artery bypass (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren (N=37) | Losartan (N=37)
Palpitations (Cardiac disorders) | 2 | 5
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Oedema peripheral (General disorders) | 3 | 0
Bronchitis (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 3
Influenza (Infections and infestations) | 1 | 4
Nasopharyngitis (Infections and infestations) | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Dizziness (Nervous system disorders) | 4 | 3
Headache (Nervous system disorders) | 4 | 6
Renal colic (Renal and urinary disorders) | 2 | 1
Hypertension (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety